CLINICAL TRIAL: NCT02370121
Title: Effect of Gymnema Sylvestre Administration on Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Brief Title: Effect of Gymnema Sylvestre on Metabolic Syndrome and Insulin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-271281-YZ
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Metabolic Syndrome
Keywords: Gymnema Sylvestre; Insulin Secretion; Insulin Sensitivity; Central Obesity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Obesity, Abdominal | interventions — Gurmarin protein, Gymnema sylvestre

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 600 mg dose per day. Two capsules of 300 mg, one in the morning with the first meal and the other at dinner during 90 days.
  Interventions: Drug: Placebo
- Gymnema Sylvestre (Experimental): 600 mg dose per day. Two capsules of 300 mg, one in the morning with the first meal and the other at dinner during 90 days.
  Interventions: Drug: Gymnema Sylvestre

INTERVENTIONS:
Drug: Placebo — Capsules of 300 mg two times per day before breakfast and dinner a total dose of 600 mg per day. During 90 days.
  Other Names: Calcined Magnesia
  Arms: Placebo
Drug: Gymnema Sylvestre — Capsules of 300 mg of calcined magnesium two times per day before breakfast and dinner a total dose of 600 mg per day. During 90 days.
  Other Names: Gurmar
  Arms: Gymnema Sylvestre

SUMMARY:
Gymnema sylvestre has demonstrated promising effects in the treatment of obesity, dyslipidemia, hypertension, insulin secretion, among others. The above mentioned findings show that Gymnema sylvestre has an excellent potential for the prevention and treatment of metabolic syndrome.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial was carried out in 24 patients with a diagnosis of metabolic syndrome in accordance with the modify International Diabetes Federation criteria. The patients received 300 mg capsules of Gymnema sylvestre or placebo, two times daily before breakfast and dinner for 90 days. Before and after intervention the investigators evaluated: The components of metabolic syndrome (waist circumference, triglycerides, high-density lipoprotein, fasting glucose and blood pressure), body weight, body mass index, total cholesterol, low-density lipoprotein, very-low-density lipoprotein, creatinine, aspartate transaminase and alanine transaminase.

Were calculated: Areas under the curve of glucose and insulin were calculated with de Trapezoidal formula. Total insulin secretion was evaluated with the Insulinogenic index and the insulin sensitivity was estimated using the Matsuda index.

ELIGIBILITY:
Inclusion Criteria:

* Letter of consent and release signed by each patient
* Body mass index: 25-34.99 kg/m2
* Body weight without variations above or under 5% during the three months prior to the study
* Diagnostic of metabolic syndrome according to the modified International Diabetes Federation definition: Central obesity (defined as waist circumference ≥ 80 cm in women and ≥ 90 cm in men)

Plus any two of the following four factors:

* Triglycerides: 150-499 mg/dL.
* High density lipoprotein: Woman < 50 mg/dL, man < 40 mg/dL.
* Blood pressure systolic:130-139 mmHg and/or Blood pressure diastolic: 85-89 mmHg
* Fasting glucose: 100-125 mg/dL

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Previous pharmacological treatment for components of metabolic syndrome
* Mental or physical illness interfering with the study
* Thyroid or cardiovascular disease
* Pregnant or suspected pregnant women
* Woman breastfeeding
* Index of body mass: ≥ 35 kg/m2
* Treatments known to affect metabolism of glucose, fats and affecting arterial tension
* Patients with hepatic or renal diseases background
* Patients diagnosed with kidneys disease
* Calcined magnesium intolerance
* Gymnema Sylvestre intolerance

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lann D, LeRoith D. Insulin resistance as the underlying cause for the metabolic syndrome. Med Clin North Am. 2007 Nov;91(6):1063-77, viii. doi: 10.1016/j.mcna.2007.06.012. PMID 17964909
- [Background] Abdul-Ghani MA, Matsuda M, Balas B, DeFronzo RA. Muscle and liver insulin resistance indexes derived from the oral glucose tolerance test. Diabetes Care. 2007 Jan;30(1):89-94. doi: 10.2337/dc06-1519. PMID 17192339
- [Background] Sandeep S, Gokulakrishnan K, Velmurugan K, Deepa M, Mohan V. Visceral & subcutaneous abdominal fat in relation to insulin resistance & metabolic syndrome in non-diabetic south Indians. Indian J Med Res. 2010 May;131:629-35. PMID 20516533
- [Result] Al-Romaiyan A, Liu B, Asare-Anane H, Maity CR, Chatterjee SK, Koley N, Biswas T, Chatterji AK, Huang GC, Amiel SA, Persaud SJ, Jones PM. A novel Gymnema sylvestre extract stimulates insulin secretion from human islets in vivo and in vitro. Phytother Res. 2010 Sep;24(9):1370-6. doi: 10.1002/ptr.3125. PMID 20812281
- [Result] Shigematsu N, Asano R, Shimosaka M, Okazaki M. Effect of administration with the extract of Gymnema sylvestre R. Br leaves on lipid metabolism in rats. Biol Pharm Bull. 2001 Jun;24(6):713-7. doi: 10.1248/bpb.24.713. PMID 11411567
- [Result] Baskaran K, Kizar Ahamath B, Radha Shanmugasundaram K, Shanmugasundaram ER. Antidiabetic effect of a leaf extract from Gymnema sylvestre in non-insulin-dependent diabetes mellitus patients. J Ethnopharmacol. 1990 Oct;30(3):295-300. doi: 10.1016/0378-8741(90)90108-6. PMID 2259217
- [Result] Porchezhian E, Dobriyal RM. An overview on the advances of Gymnema sylvestre: chemistry, pharmacology and patents. Pharmazie. 2003 Jan;58(1):5-12. PMID 12622244
- [Result] Koshu K, Hirota S, Sonobe M, Takahashi S, Takaku A, Saito T, Ushijima T. [Continuous recording of cerebral blood flow by means of thermal diffusion method using Peltier stack]. Neurol Med Chir (Tokyo). 1987 Aug;27(8):724-8. doi: 10.2176/nmc.27.724. No abstract available. Japanese. PMID 2451154
- [Result] Bhansali S, Shafiq N, Pandhi P, Singh AP, Singh I, Singh PK, Sharma S, Malhotra S. Effect of a deacyl gymnemic acid on glucose homeostasis & metabolic parameters in a rat model of metabolic syndrome. Indian J Med Res. 2013 Jun;137(6):1174-9. PMID 23852298
- [Result] Tiwari P, Mishra BN, Sangwan NS. Phytochemical and pharmacological properties of Gymnema sylvestre: an important medicinal plant. Biomed Res Int. 2014;2014:830285. doi: 10.1155/2014/830285. Epub 2014 Jan 6. PMID 24511547
- [Result] Kumar V, Bhandari U, Tripathi CD, Khanna G. Protective Effect of Gymnema sylvestre Ethanol Extract on High Fat Diet-induced Obese Diabetic Wistar Rats. Indian J Pharm Sci. 2014 Jul;76(4):315-22. PMID 25284929
- [Result] Astell KJ, Mathai ML, Su XQ. Plant extracts with appetite suppressing properties for body weight control: a systematic review of double blind randomized controlled clinical trials. Complement Ther Med. 2013 Aug;21(4):407-16. doi: 10.1016/j.ctim.2013.05.007. Epub 2013 Jun 24. PMID 23876572
- [Result] Al-Romaiyan A, King AJ, Persaud SJ, Jones PM. A novel extract of Gymnema sylvestre improves glucose tolerance in vivo and stimulates insulin secretion and synthesis in vitro. Phytother Res. 2013 Jul;27(7):1006-11. doi: 10.1002/ptr.4815. Epub 2012 Aug 21. PMID 22911568
- [Result] Ogawa Y, Sekita K, Umemura T, Saito M, Ono A, Kawasaki Y, Uchida O, Matsushima Y, Inoue T, Kanno J. [Gymnema sylvestre leaf extract: a 52-week dietary toxicity study in Wistar rats]. Shokuhin Eiseigaku Zasshi. 2004 Feb;45(1):8-18. doi: 10.3358/shokueishi.45.8. Japanese. PMID 15168555
- [Result] Okabayashi Y, Tani S, Fujisawa T, Koide M, Hasegawa H, Nakamura T, Fujii M, Otsuki M. Effect of Gymnema sylvestre, R.Br. on glucose homeostasis in rats. Diabetes Res Clin Pract. 1990 May-Jun;9(2):143-8. doi: 10.1016/0168-8227(90)90106-4. PMID 1695875
- [Result] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Result] Tai MM. A mathematical model for the determination of total area under glucose tolerance and other metabolic curves. Diabetes Care. 1994 Feb;17(2):152-4. doi: 10.2337/diacare.17.2.152. PMID 8137688
- [Result] Renga B, Festa C, De Marino S, Di Micco S, D'Auria MV, Bifulco G, Fiorucci S, Zampella A. Molecular decodification of gymnemic acids from Gymnema sylvestre. Discovery of a new class of liver X receptor antagonists. Steroids. 2015 Apr;96:121-31. doi: 10.1016/j.steroids.2015.01.024. Epub 2015 Feb 7. PMID 25668616
- [Result] Stumvoll M, Mitrakou A, Pimenta W, Jenssen T, Yki-Jarvinen H, Van Haeften T, Renn W, Gerich J. Use of the oral glucose tolerance test to assess insulin release and insulin sensitivity. Diabetes Care. 2000 Mar;23(3):295-301. doi: 10.2337/diacare.23.3.295. PMID 10868854
- [Result] Izutani Y, Murai T, Imoto T, Ohnishi M, Oda M, Ishijima S. Gymnemic acids inhibit rabbit glyceraldehyde-3-phosphate dehydrogenase and induce a smearing of its electrophoretic band and dephosphorylation. FEBS Lett. 2005 Aug 15;579(20):4333-6. doi: 10.1016/j.febslet.2005.06.070. PMID 16054141
- [Result] Wang Y, Dawid C, Kottra G, Daniel H, Hofmann T. Gymnemic acids inhibit sodium-dependent glucose transporter 1. J Agric Food Chem. 2014 Jun 25;62(25):5925-31. doi: 10.1021/jf501766u. Epub 2014 Jun 10. PMID 24856809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Gymnema Sylvestre
Started | 12 | 12
Completed | 11 (One patient did not complete the study due to early withdrawl) | 11 (One patient did not complete the study due to early withdrawl)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gymnema Sylvestre | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (4) | 43 (1) | 42 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Body weight (BW) [Mean (Standard Deviation); unit: kg] — The BW was evaluated after an overnight fast, through a bioimpedance digital scale results are reported in kilograms with a decimal.
  kg | 78.8 (16.1) | 81.3 (10.6) | 80.2 (15.4)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — The BMI was calculated by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
  kg/m^2 | 30.29 (3.21) | 31.24 (2.55) | 30.56 (2.98)
Waist circumference (WC) [Mean (Standard Deviation); unit: cm] — The WC was evaluated after an overnight fast with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  cm | 98 (14) | 99 (10) | 98 (14)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — The SBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of SBP. The value was expressed on mmHg.
  mmHg | 123 (11) | 121 (10) | 122 (15)
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — The DBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of DBP. The value was expressed on mmHg.
  mmHg | 81 (7) | 79 (5) | 81 (6)
Triglycerides (TGs) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of TGs, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 2.91 (0.93) | 2.37 (1.03) | 2.69 (0.90)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of TC, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 4.53 (0.52) | 4.60 (1.06) | 4.59 (0.63)
high-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of HDL-C, was taken after an overnight fast and was evaluated by colorimetric method. The value was expressed on mmol/L.
  mmol/L | 1.00 (0.23) | 1.11 (0.18) | 1.04 (0.22)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of LDL-C, was taken after an overnight fast and was calculated by Friedewald formula. The value was expressed on mmol/L.
  mmol/L | 2.12 (0.59) | 2.48 (0.93) | 2.15 (0.52)
Very-low density lipoprotein (VLDL) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining the VLDL, was taken after an overnight fast and was calculated as triglycerides/5 . The value was expressed on mmol/L.
  mmol/L | 0.54 (0.17) | 0.45 (0.15) | 0.49 (0.16)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of FPG, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 4.97 (0.44) | 5.22 (0.72) | 5.09 (0.58)
2-hour postload plasma glucose (2-h PG) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of 2-h PG, was taken two hours after the ingestion of the drink with 75 g dextrose and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 7.72 (1.78) | 7.61 (1.89) | 7.67 (184)
Area under the curve of glucose (AUCG) [Mean (Standard Deviation); unit: mmol/L/min] — The estimation for AUCG was calculated from parameters obtained during the 2 hours oral glucose tolerant test (OGTT) with 75 g dextrose by trapezoidal integration. The value was expressed mmol/L/min.
  mmol/L/min | 972 (154) | 979 (182) | 976 (168)
Area under the curve of insulin (AUCI) [Mean (Standard Deviation); unit: pmol/L/min] — The estimation for AUCI was calculated from parameters obtained during the 2 hours oral glucose tolerant test (OGTT) with 75 g dextrose by trapezoidal integration. The value was expressed on pmol/L/min.
  pmol/L/min | 64314 (34914) | 61626 (29700) | 62970 (32307)
Total insulin secretion [Mean (Standard Deviation); unit: unitless] — Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin / ΔABC glucose).
  unitless | 0.61 (0.33) | 0.57 (0.24) | 0.59 (0.57)
First phase of insulin secretion [Mean (Standard Deviation); unit: unitless] — First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0').
  unitless | 1403 (682) | 1458 (510) | 1431 (596)
Insulin sensitivity [Mean (Standard Deviation); unit: unitless] — Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)].
  unitless | 3.3 (1.9) | 3.8 (1.1) | 3.6 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Waist Circumference (WC)
Description: The WC was evaluated after an overnight fast with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
Time Frame: Week 12
Population: All participants, including those who dropped out before the end were taken into account for statical analysis (intention to treat).
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
cm | 101 (15) | 96 (7)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Triglycerides (TGs)
Description: The blood sample for determining of TGs, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L | 2.79 (0.59) | 1.70 (0.75)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

3. Primary Outcome: High-density Lipoprotein Cholesterol (HDL-C)
Description: The blood sample for determining of HDL-C, was taken after an overnight fast and was evaluated by colorimetric method. The value was expressed on mmol/L.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L | 1.03 (0.25) | 1.08 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Fasting Plasma Glucose (FPG)
Description: The blood sample for determining of FPG, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L | 5.00 (0.61) | 4.83 (0.72)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Systolic Blood Pressure (SBP)
Description: The SBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of SBP. The value was expressed on mmHg.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmHg | 122 (13) | 121 (11)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Diastolic Blood Pressure (DBP)
Description: The DBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of DBP. The value was expressed on mmHg.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmHg | 83 (7) | 78 (8)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Total Insulin Secretion
Description: The total insulin secretion was calculated by the insulinogenic index (ΔABC insulin / ΔABC glucose).
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
unitless | 0.95 (0.66) | 0.59 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney)

8. Primary Outcome: First Phase of Insulin Secretion
Description: The first phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0').
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
unitless | 1805 (721) | 1366 (472)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.77, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Insulin Sensitivity
Description: The insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)].
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
unitless | 2.5 (1.4) | 4.1 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Body Weight (BW)
Description: The BW was evaluated after an overnight fast, through a bioimpedance digital scale results are reported in kilograms with a decimal.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
kg | 80.3 (18.2) | 77.9 (8.4)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Body Mass Index (BMI)
Description: The BMI was calculated by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
kg/m^2 | 30.70 (3.75) | 30.43 (2.23)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Total Cholesterol (TC)
Description: The blood sample for determining of TC, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L | 5.04 (0.62) | 4.55 (0.98)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Low-density Lipoprotein Cholesterol (LDL-C)
Description: The blood sample for determining of LDL-C, was taken after an overnight fast and was calculated by Friedewald formula. The value was expressed on mmol/L.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L | 2.77 (0.54) | 2.69 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Very-low Density Lipoprotein (VLDL)
Description: The blood sample for determining the VLDL, was taken after an overnight fast and was calculated as triglycerides/5. The value was expressed on mmol/L.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L | 0.56 (0.12) | 0.35 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: 2-hour Postload Plasma Glucose (2-h PG)
Description: The blood sample for determining of 2-h PG, was taken two hours after the ingestion of the drink with 75 g dextrose and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L | 6.83 (2.00) | 7.22 (3.05)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Area Under the Curve of Glucose (AUCG)
Description: The estimation for AUCG was calculated from parameters obtained during the 2 hours oral glucose tolerant test (OGTT) with 75 g dextrose by trapezoidal integration. The value was expressed mmol/L/min.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: mmol/L/min
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
mmol/L/min | 965 (235) | 914 (267)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Area Under the Curve of Insulin (AUCI)
Description: The estimation for AUCI was calculated from parameters obtained during the 2 hours oral glucose tolerant test (OGTT) with 75 g dextrose by trapezoidal integration. The value was expressed on pmol/L/min.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: pmol/L/min
Arm/Group | Placebo | Gymnema Sylvestre
Number analyzed (Participants) | 11 | 11
pmol/L/min | 90816 (45336) | 60468 (37290)
Statistical Analysis 1: Comparison: Placebo vs Gymnema Sylvestre; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 90 days of the study.
Arm/Group | Placebo | Gymnema Sylvestre
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Gymnema Sylvestre (N=12)
headache (Nervous system disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No